CLINICAL TRIAL: NCT06652802
Title: Effectiveness of Nurse-Conducted Brief Intervention (NCBI) Supplemented With Mobile-based Application for Monitoring and Relapse Prevention in Patients With Alcohol Use Disorders: A Randomized Controlled Trial
Brief Title: Effectiveness of Nurse-Conducted Brief Intervention (NCBI) Supplemented With Mobile for Preventing Alcohol Use Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor of Psychiatry and Human Genetics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23090050; 5D43TW009114-10 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Use Disorders (AUDs),; A Randomized controlled trial; Gastroenterology,; CIWA,; Nurse-Conducted Brief Intervention (NCBI)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: The study design is a randomized controlled trial. In this type of study, participants are randomly assigned to two different groups, i.e Group A and Group B.
  Group A participants receive only Nurse-Conducted Brief Intervention (NCBI). Whereas's Group B receives Nurse-Conducted Brief Intervention (NCBI). supplemented with mobile based application.
  The study is designed as single-blind, meaning the outcome assessors and the data analysts will be blinded to the group allocations to reduce bias in the evaluation of the outcomes
Who Masked: Outcomes Assessor
Masking Description: The study is designed as single-blind, meaning the outcome assessors and the data analysts will be blinded to the group allocations to reduce bias in the evaluation of the outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Conducted Brief Intervention (NCBI). supplemented with mobile based application (Experimental): Experimental group participants receive Nurse-Conducted Brief Intervention (NCBI). supplemented with mobile based application. Due to the availability of Nurse Conducted Brief intervention (NCBI) service in Gastroenterology department by trained nurse it was done in the gastroentrology department.
  Interventions: Behavioral: Nurse-Conducted Brief Intervention (NCBI). supplemented with mobile based application.
- Nurse-Conducted Brief Intervention (NCBI) (Active Comparator): Control group participants receive only Nurse-Conducted Brief Intervention (NCBI).
  Interventions: Behavioral: Nurse-Conducted Brief Intervention (NCBI)

INTERVENTIONS:
Behavioral: Nurse-Conducted Brief Intervention (NCBI). supplemented with mobile based application. — * An interactive mobile based application will be developed with the following features to assist in monitoring and preventing relapse.
  * Purpose of the Mobile based application: The mobile application will be an interactive tool designed to assist in monitoring and preventing relapse of alcohol use disorder. It will provide various features to support users in their journey to sobriety, including personalized recovery plans, goal setting, progress tracking, stress and craving management tools, educational resources, daily reflection prompts, emergency assistance, personalized reminders, progress reports, and psychoeducational videos.
  * The Target population: 40 Male patients selected through randomized sampling, aged between 18 and 59 years, who have participated in Nurse-Conducted Brief Intervention (NCBI) for AUD in the Gastroenterology ward with diagnosis of alcohol dependence use disorder based on ICD-10 who have access to smartphone application and have the ability to use it.
  Arms: Nurse-Conducted Brief Intervention (NCBI). supplemented with mobile based application
Behavioral: Nurse-Conducted Brief Intervention (NCBI) — * Nurse-Conducted Brief Intervention (NCBI) is a feasible and acceptable model of care for males diagnosed with Alcohol Use Disorders (AUDs) in gastroenterology settings. The study found that the Nurse-Conducted Brief Intervention (NCBI) had a positive impact on promoting abstinence in patients with AUDs, and the preliminary findings demonstrate probable good outcomes. [21].
  * It consists of a trained Nurse delivering three individual sessions with the patient over a span of two to three days (15 to 20 mins each) during their period of admission in the ward and one session with the family members.
  Arms: Nurse-Conducted Brief Intervention (NCBI)

SUMMARY:
The study is aimed to find out that combining Nurse-Conducted Brief Intervention (NCBI) with a Smart Mobile is better than Nurse-Conducted Brief Intervention (NCBI) only in preventing relapse among Alcohol Use Disorder patients. The high relapse rates among alcohol disorder patients may be benefitted by new technology using application for improved outcomes in managing and preventing alcohol addiction relapse.

DETAILED DESCRIPTION:
A Meta-analysis including 34 studies showed that Brief Intervention helped in reducing the amount of alcohol consumption after a study duration of 1 year in comparison with the control group. In India, there have been few studies on Brief Intervention. A comparison study of Brief intervention versus simple advice for Alcohol Use Disorder was conducted in North India in 2007, which showed a slight advantage for Brief intervention. But the results were not showing a significant outcome and it was concluded that booster sessions were required. A review of literature revealed that comprehensive recovery management systems using the capabilities of smart-phones to provide a variety of tools and services that can be tailored to individuals, including in-the-moment assessments and access to peer discussion groups have the strongest theoretical base and have yielded the strongest and longest-lasting effects for management of alcohol use disorders. [10]. A study review revealed that smartphone application has the potential to monitor alcohol use and craving in the natural environment and deliver tailored treatment to users when they need it most. A study revealed that smartphone-delivered coping strategies for alcohol cravings are effective in reducing craving cued drinking and that craving cues related to drinking environments and drinking times of day represent fruitful areas of intervention focus.

JUSTIFICATION / NEED FOR THE STUDY The present studies suggest that a substantial proportion of patients with alcohol use disorders relapse to alcohol during the course of treatment. Efforts are required to delay and avoid such relapse and maintain abstinence by effective treatment approaches. A major barrier to care is the lack of adequately skilled human resources to deliver contextually appropriate treatments. Nurse-conducted Brief Intervention supplemented with mobile application-based can be a beneficial approach to prevent relapse and support patients in their journey to overcome alcohol addiction. It also promotes a more continuous and connected recovery process by enabling regular communication and data sharing between the user and their counsellor.

Proposed Methodology: Only males will be included in the study.

* Including women in this study would necessitate a gender-specific analysis [5], which could complicate the primary objective of evaluating the combined intervention of Nurse-Conducted Brief Intervention (NCBI) and a mobile based application.
* To maintain the internal validity of this study and to ensure a clear, focused evaluation of the intervention, the investigators have chosen to initially focus on male participants.
* The non-availability of female patients or a smaller number of female patients according to hospital admission records diagnosed with alcohol dependence admitted to the hospital ward due to stigma will also affect the data collection process.
* Future studies will aim to address the effectiveness of these interventions specifically for women, considering their unique needs and responses to treatment.

SAMPLE SIZE and the BASIS for the same:

The sample size was calculated using the Sample size calculator (riskcalc.org) for superiority trial with a dichotomous outcome. The investigators based the analysis on the prevalence rates of 65% by a study in Bangalore, with a 2-side significance level of 0.05, Power (1-beta) of 0.8, Ratio of sample size (unexposed/exposed) of 1, Probability of event in the unexposed group =0.6, Probability of event in the exposed group = 0.4, margin of difference of 0.5, with a 10% dropout rate, the sample size estimated was 74 (34 in each group).

Considering the drop out, approximately 40 patients will be taken in each group to achieve the target recruitment.

Study design: A Randomized controlled trial Study site: In-patient setting of Department of Gastroenterology, St John's Medical College, Bangalore.

Reasons for the recruitment of subjects from the Gastroenterology department:

* Due to the availability of Nurse Conducted Brief intervention (NCBI) service in Gastroenterology department by trained nurse.
* High prevalence of Alcohol Use Disorders (AUDs) among patients admitted in Gastroenterology department. Patients in this unit often present with issues directly related to their alcohol use, making it an ideal setting for intervention.
* Subjects who are not currently in withdrawal and have been deemed medically stable by the treating physician in the Gastroenterology unit will be enrolled for the study. This ensures that participants are medically stable and suitable for the study.

Study Period: 1 year Method of sampling: Randomized sampling, the study design is a randomized controlled trial. In this type of study, participants are randomly assigned to two different groups, i.e STATISTICAL ANALYSIS The data will be reviewed for normality. The data will be presented as parametric or non- parametric depending on the distribution. The chi-squared test will be used to find the difference between categorical variables. An Independent sample t test would be used to find the differences between the means of the two groups. Repeated measure ANOVA will be used for the outcome measures.

ETHICAL CONSIDERATION

* The study will commence after IEC approval (SJMC) and IRB approval of protocol of the study.
* Confidentiality will be maintained.
* Participation will be voluntary Approval of the Institutional Ethics committee will be sought. Permission from the Head of Department of Gastroenterology will be sought to enrol patients from the department of Gastroenterology. The participants will be briefed on the study and provided with explanations on how the gathered medical data could be used. Informed consent will be obtained from the patients prior to enrolling in the study.

Screening:

* All patients with alcohol use disorder will be identified through inclusion and exclusion criteria from inpatient settings of the Gastroenterology department at SJMCH. Confidentiality will be maintained.
* They will be assessed with the Clinical Institute Withdrawal Assessment of Alcohol Scale, revised (CIWA-Ar) for monitoring withdrawal symptoms.
* CIWA-Ar score less than 8 or after 3 days of admission the patient will be screened for major psychiatric illness using Modified Mini Screen (MMS).
* The Modified Mini Screen (MMS) is a generic screening measure for mood, anxiety, and psychotic spectrum disorders. There are twenty-two questions with yes/no responses. It takes about fifteen minutes to complete.

Baseline Assessment:

* The Socio-demographic details will be collected from participants using BIG proforma.
* Brief Intervention in Gastroenterology proforma is an initiative of the Department of Psychiatry, St. John's Medical College, Bangalore, which includes informed consent, socio-demographic details of the participants, details regarding their drinking pattern, LFT values, 4 sessions of Brief Intervention and follow up status (abstinent, lapse, relapse, expired).
* The Severity of Alcohol Dependence Questionnaire (SADQ) will be used to assess the severity of alcohol dependence. Severity of Alcohol Dependence Questionnaire (SADQ) is a short, easy-to-complete, self-administered, 20-item questionnaire designed to measure severity of dependence on alcohol.
* Alcohol Use Disorder Identification Test questionnaire will be used to screen the patient for alcohol use disorders. The Alcohol Use Disorders Identification Test [AUDIT] is a 10-item screening tool developed by the World Health Organization [WHO] to assess alcohol consumption, drinking behaviours, and alcohol-related problems. The AUDIT has been validated across genders and in a wide range of racial/ethnic groups and is well suited for use in primary care settings. Scores for each question range from 0-4. For questions 9 and 10, which only have three responses, the scoring is 0, 2 and 4 [from left to right]. A score of 8 or more is associated with harmful or hazardous drinking
* Readiness to change questionnaire will be used to assess the motivation to abstain from alcohol. This questionnaire is used to assess how they are motivated to abstain from alcohol. It has 12 questions and is scored from -2 to 2, -2 being strongly disagree, -1(disagree), 0(unsure), 1(agree), 2(strongly agree).
* The whole study is a three-time assessment which might take approximately 30- 40 minutes to assess.
* It will be ensured that the caregiver is not made to travel exclusively for the purpose of this study.

  * MMS: Modified Mini Screen
  * CIWA - Ar: Clinical Institute Withdrawal Assessment of Alcohol Scale, revised
  * BIG-P: Brief Intervention in Gastroenterology Proforma
  * SADQ: The Severity of Alcohol Dependence Questionnaire
  * AUDIT: Alcohol Use Disorder Identification Test questionnaire
  * RTC-TRV: Readiness to Change Questionnaire

Follow-up

Follow-Up Details: 1-Month and 3-Month Follow-Ups:

Querying on alcohol use will occur during these follow-ups. Follow up assessment will be done virtually with telephonic phone calls.

1. 1-Month Follow-Up: After 1 month of enrolment, participants from both groups will be followed up by the research team through telephonic phone call. Follow-up assessments include outcomes like relapse, lapse, or maintaining abstinence along with use of assessment tools like SADQ, AUDIT, and readiness to change.
2. 3-Month Follow-Up: Like the 1-month follow-up, participants from both groups will undergo follow-up assessments after 3 months.

   * In addition to Follow up assessment done virtually with telephonic phone calls, daily tracking in the mobile based application will be used as an additional source of information regarding the abstinence and relapse use of alcohol by the participant with the consent of participant.
   * Participants randomized to the mobile health application group are expected to continue using the mobile health application regularly after discharge from the hospital.
   * It is highly encouraged that the mobile health application is used at least once daily to track the progress, utilize its features, and receive ongoing support for a minimum period of 3 months.
   * This regular usage is a crucial part of the study, and participants are encouraged to engage with the mobile health application up to the 3-month follow-up point to maximize the intervention's benefits

The follow-up assessment will be done using following:

* Brief Intervention in Gastroenterology Proforma (BIG- P)
* The Severity of Alcohol Dependence Questionnaire (SADQ)
* Alcohol Use Disorder Identification Test questionnaire (AUDIT)
* Readiness to Change Questionnaire (RTC -TRV)

ELIGIBILITY:
Inclusion Criteria:

* Male patients.
* Aged between 18 and 59 years.
* Diagnosis of alcohol dependence use disorder based on ICD-10 criteria.
* Patients with an Android smartphone and the ability to use mobile application.

Exclusion Criteria:

* Female patients
* Comorbid other substance abuse, except tobacco.
* Comorbid major mental illness /physical illness.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — • Female patients were excluded from the study. The decision to exclude women from the study is likely grounded in the consideration of potential gender-specific factors in the manifestation and treatment of Alcohol Use Disorders (AUDs). Research suggests that there are gender differences in the prevalence, patterns, and consequences of alcohol consumption, as well as in the response to interventions for alcohol-related issues, which will affect the outcome of the study.
Enrollment: 74 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Nurse-Conducted Brief Intervention (NCBI) supplemented with a Mobile Health Application in preventing relapse among patients with Alcohol Use Disorders (AUDs | Three months period
  The primary endpoint of the study is the effectiveness of Nurse-Conducted Brief Intervention (NCBI) supplemented with a Mobile Health Application in preventing relapse among patients with Alcohol Use Disorders (AUDs) over a three-month period.
  • The primary outcome measure will be the difference in relapse rates between the group receiving NCBI with the mobile application and the group receiving only NCBI.

SECONDARY OUTCOMES:
Provide insight into the effectiveness and impact of the interventions: Sociodemographic | Baseline
  Assessment of socio-demographic factors, such as age, gender, education, and occupation, and their association with relapse.
Provide insight into the effectiveness and impact of the interventions: Severity of AUD | Baseline
  Evaluation of the severity of Alcohol Use Disorder using standardized assessment tools like the Severity of Alcohol Dependence Questionnaire (SADQ).A score of 31 or higher indicates "severe alcohol dependence".A score of 16 -30 indicates "moderate dependence".A score of below 16 usually indicates only a mild physical dependency.
  A score of 16 -30 indicates "moderate dependence"
Provide insight into the effectiveness and impact of the interventions:Lapse evaluation | Baseline
  Examination of the secondary outcome measures, including Lapse (occasional drinking without significant impairment), Abstinence (complete avoidance of alcohol), and Relapse (return to heavy drinking after a period of abstinence).
Provide insight into the effectiveness and impact of the interventions: comparison with sociodemographic factors | Baseline
  Comparison of the secondary outcome measures with socio-demographic factors and severity of AUD to understand potential predictors of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh

IPD SHARING:
Plan to Share IPD: Yes
* Strategic measures have been diligently put in place to safeguard the confidentiality and privacy of participants' data. .
  * Data that is shared with external collaborators is meticulously stripped of any personal identifiers, rendering it completely de-identified and anonymized.
  * Any external sharing of data will be conducted under an approved Data Use Agreement (DUA) to ensure compliance with ethical and privacy standards. Should the need arise for scientific analysis or the creation of research papers, only this de-identified data will be shared with external collaborators. This selective sharing of information strikes a delicate balance between scientific collaboration and ethical responsibility.
  * By sharing data that has been meticulously stripped of any potential identifying markers, the research maintains the integrity of participant anonymity while allowing for robust scientific exploration.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year
Access Criteria: The study should be ethically approved and scientifically sound,